CLINICAL TRIAL: NCT00504465
Title: Cervical Ripening and Induction of Labor: a Randomized Controlled Trial of Combined Versus Sequential Use of Dinoprostone and Oxytocin.
Brief Title: Combined Agent Randomized Trial of Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0402-264
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Labor Induction; Cervical Ripening
Keywords: Labor; Labor induction; Cervical ripening; Dinoprostone; Fetal safety; Oxytocin; Cesarean delivery
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dinoprostone

SUMMARY:
To compare sequential dinoprostone and oxytocin for induction of labor at term with intact membranes and an unripe cervix to two simultaneous regimens. Our aim was to confirm findings from smaller trials and add to data on fetal safety.

DETAILED DESCRIPTION:
This study is a non-blinded, three arm randomized trial at 3 sites. Entry criteria were: >36 weeks' singleton, cephalic gestation with intact membranes and an unripe cervix (Bishop's score <6). Study arms were: 1) dinoprostone vaginal insert (Cervidil) for 12 hours followed by oxytocin, 2) dinoprostone vaginal insert (Cervidil) for 12 hours with simultaneous oxytocin, and 3) intracervical dinoprostone gel (Prepidil)(one dose) followed by immediate oxytocin. Primary outcome measure was the rate of vaginal delivery <24 hours. Secondary outcomes were randomization to delivery interval, rate of cesarean delivery (CD) for non reassuring fetal status (NRFS) and rate of uterine hyperstimulation.

ELIGIBILITY:
Inclusion Criteria:

* > or = to 36 weeks of gestation
* Singleton fetus
* Cephalic presentation
* Intact membranes and an unripe cervix (Bishop score <6)

Exclusion Criteria:

* Multifetal gestation
* Rupture of membranes
* Ripe cervix (Bishop score >6)
* Active labor
* Contraindication to vaginal delivery
* Previous uterine surgery
* Non-cephalic presentation
* Fetal macrosomia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210
Dates: Start 2002-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Rate of vaginal delivery <24 hours

SECONDARY OUTCOMES:
Randomization to delivery interval
Rate of cesarean delivery for non reassuring fetal status
Rate of uterine hyperstimulation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Skupski, MD, Principal Investigator — Weill Medical College of Cornell University; Michael Cabbad, MD, Principal Investigator — The Brooklyn Hospital Center
Locations (3):
- United States (3):
  - The Brooklyn Hospital Center, Brooklyn, New York
  - New York Hospital Medical Center of Queens, Flushing, New York
  - Weill Medical College of Cornell University, New York, New York